CLINICAL TRIAL: NCT02026921
Title: A Phase II Study of Docetaxel and Carboplatin as Second Line Chemotherapy in First Relapse of Platinum Sensitive Epithelial Ovarian Cancer
Brief Title: A Phase II Study of Docetaxel and Carboplatin in Late Relapse of Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSGO-OC-0303
Record Dates: First submitted 2013-12-18; First posted 2014-01-03 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2013-12

CONDITIONS: Ovarian Epithelial Cancer Recurrent
Keywords: Phase II study,; Recurrent platinum-sensitive ovarian cancer; docetaxel; Carboplatin; Toxicity
MeSH Terms: interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin and docetaxel (Experimental): Intravenous infusion every 3 weeks Carboplatin plus docetaxel
  Interventions: Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Carboplatin — Carboplatin, AUC5, IV (in the vein) on day 1 of each 21 day cycle. Number of Cycles: 6 or until progression or unacceptable toxicity develops
Drug: Docetaxel — 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle. Number of Cycles: 6 or until progression or unacceptable toxicity develops.
  Other Names: Taxotere

SUMMARY:
A phase II single arm study of carboplatin and docetaxel in treatment of first sensitive relapse of epithelial ovarian, peritoneal or tubal cancer.

Hypothesis: Treatment with this combination in second line is safe and with a low frequency of neurologic side effect.

DETAILED DESCRIPTION:
Evaluation of toxicity and response of treatment with carboplatin and docetaxel to patients with epithelial cancer of ovary, fallopian tube or peritoneum with their first relapse occurring at least 6 months after end of first line treatment- Evaluation of toxicity according to Clinical Toxicity Criteria version 2.

ELIGIBILITY:
Inclusion Criteria:

* Epithelial carcinoma of ovarian, peritoneal or fallopian tube origin.
* Female
* age above 18 years
* WHO performance status 0-2
* Life expectancy > 3 months
* Previous treatment with one platinum and taxane containing regimen.
* Platinum and taxane sensitive relapse
* At least one evaluable/measurable lesion.
* Adequate hematologic, renal and liver function
* Consent form signed and dated before inclusion

Exclusion Criteria:

* Prior treatment with more than one line of chemotherapy
* Concurrent severe and/or uncontrolled co-morbid medical condition.
* History of previous or concurrent malignancy within the previous 5 years • History of prior serious allergic reactions such as anaphylactic shock
* Pregnant or lactating women (or potentially fertile women not using adequate contraception)
* Peripheral neuropathy > Grade 2
* History of allergy to drugs containing the excipient TWEEN 80®.
* Concomitant administration of any other experimental drug under investigation or concurrent treatment with any other anti-cancer therapy
* Clinical evidence of brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 30 days after last chemotherapy course
  Safety will be established by grading the observed toxicities using the NCI Common Toxicity Criteria (CTC Version 2.0). All toxicities observed within 30 dayes of last chemocourse will be included.

SECONDARY OUTCOMES:
Response rate | Up to 30 dayes after last chemotherapy course
  Response rate according to Resist 1.0 Response rate is the proportion of patients that achieve CR or PR.
Progression free survival | Up to 3 year
  Time from start of treatment to the earlier date of assessment of progression or death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar B Kristensen, MD, PhD, Study Chair — NSGO-CTU
Locations (4):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Herlev University Hospital, Copenhagen
- Tampere University Hospital, Tampere, Finland
- Norwegian Radium Hospital, Oslo, Norway